CLINICAL TRIAL: NCT05119790
Title: An Open Label, Phase 1 Study of Mass Balance, Pharmacokinetics, Metabolite Profile, and Metabolite Identification of a Single Oral Dose of [14C]-BIIB122 ([14C] DNL151) in Healthy Male Subjects
Brief Title: A Study of Mass Balance, Pharmacokinetics, Metabolite Profile, and Metabolite Identification of BIIB122/DNL151 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: Denali Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 283HV102
Record Dates: First submitted 2021-08-27; First posted 2021-11-15 (Actual); Last update posted 2021-12-07 (Actual); Status verified 2021-11

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — DNL151

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cohort A (Experimental)
  Interventions: Drug: [14C] BIIB122 ([14C] DNL151)

INTERVENTIONS:
Drug: [14C] BIIB122 ([14C] DNL151) — Oral dose

SUMMARY:
This is a single-center, non-randomized, open-label Phase 1 study to determine the absorption, metabolism, and excretion (AME) of BIIB122 (DNL151) following administration of a single oral dose of [14C] BIIB122 ([14C] DNL151) following a fast. The mass balance, excretion, and PK of BIIB122 (DNL151) will be used to evaluate AME.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4)(A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
key Inclusion Criteria:

* For men who choose to have sex with women, either: vasectomy, use of condoms, or sex with a woman who is of non-childbearing potential
* Body mass index ≥18.0 kg/m2 and ≤32.0 kg/m2
* Body weight ≥5.0 kg and ≤100.0 kg
* Considered to be in good health
* Non-smoker

Key Exclusion Criteria:

* History or presence of any condition or prior surgery that, in the opinion of the investigator, poses a significant risk to subject safety and/or achievement of study objectives

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-08-27 (Actual); Primary Completion 2021-11-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Mass balance (total recovery) following oral administration of a single dose of [14C] BIIB122 ([14C]-DNL151) | 43 days
Percentage of radioactivity recovered in urine following oral administration of a single dose of [14C] BIIB122 ([14C]-DNL151) | 43 days
Percentage of radioactivity recovered in feces following oral administration of a single dose of [14C] BIIB122 ([14C]-DNL151) | 43 days
PK Parameter: The first time to maximum observed concentration (Tmax) for total radioactivity and BIIB122 (DNL151) in blood following oral administration of a single dose of [14C]-BIIB122 ([14C]-DNL151) | 43 days
PK Parameter: Maximum observed plasma concentration (Cmax) occurring at Tmax for total radioactivity and BIIB122 (DNL151) in blood following oral administration of a single dose of [14C]-BIIB122 ([14C]-DNL151) | 43 days
PK Parameter: Area under the concentration-time curve (AUC) of total radioactivity and BIIB122 (DNL151) in blood following oral administration of a single dose of [14C]-BIIB122 ([14C]-DNL151) | 43 days
PK Parameter: Time at which half the drug has been eliminated (T1/2) of total radioactivity and BIIB122 (DNL151) in blood following oral administration of a single dose of [14C]-BIIB122 ([14C]-DNL151) | 43 days
PK Parameter: Apparent systemic clearance (CL/F) of total radioactivity and BIIB122 (DNL151) in blood following oral administration of a single dose of [14C] BIIB122 ([14C]-DNL151) | 43 days
PK Parameter: Apparent volume of distribution (Vz/F) of total reactivity and BIIB122 (DNL151) in blood following oral administration of a single dose of [14C] BIIB122 ([14C]-DNL151) | 43 days
Profiles of [14C] BIIB122 ([14C]-DNL151) and its [14C] metabolites in plasma, urine, and feces following oral administration of a single dose of [14C] BIIB122 ([14C]-DNL151) | 43 days

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | 43 days
PK Parameter: The ratio of total radioactivity in whole blood to that in plasma following oral administration of a single dose of [14C] BIIB122 ([14C]-DNL151) | 43 days
Chemical identities of the [14C] metabolites of [14C] BIIB122 ([14C]-DNL151) measured in plasma, urine, and feces | 43 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Denali Therapeutics Inc.
Locations (1):
- Pharmaron CPC, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No